#### MEDICAL RECORD

#### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

Adult Patient or

• Parent, for Minor Patient

INSTITUTE: National Cancer Institute

STUDY NUMBER: 09-C-0065 PRINCIPAL INVESTIGATOR: Wyndham Wilson, M.D., Ph.D

STUDY TITLE: Phase 1 Trial of Siplizumab and Dose-Adjusted EPOCH-Rituximab in T and NK-Cell

Lymphomas

Continuing Review Approved by the IRB on 02/05/18

Amendment Approved by the IRB on 12/18/18 (H)

Date posted to web: 12/28/18

Standard

#### INTRODUCTION

We invite you to take part in a research study at the National Institutes of Health (NIH).

First, we want you to know that:

Taking part in NIH research is entirely voluntary.

You may choose not to take part, or you may withdraw from the study at any time. In either case, you will not lose any benefits to which you are otherwise entitled. However, to receive care at the NIH, you must be taking part in a study or be under evaluation for study participation.

You may receive no benefit from taking part. The research may give us knowledge that may help people in the future.

Second, some people have personal, religious or ethical beliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). If you have such beliefs, please discuss them with your NIH doctors or research team before you agree to the study.

Now we will describe this research study. Before you decide to take part, please take as much time as you need to ask any questions and discuss this study with anyone at NIH, or with family, friends or your personal physician or other health professional.

#### Why are you being asked to take part in this study?

Lymphoma and its treatment: You have a disease called T-cell or NK cell non-Hodgkin's lymphoma which your doctors think would be best treated with chemotherapy. In general, mature T-cell and NK cell lymphomas are generally responsive to chemotherapy but less likely to be cured than B-cell lymphomas. This protocol is specifically for people with T-cell and NK cell lymphomas, as we are trying to find better treatments for these types of lymphoma.

PATIENT IDENTIFICATION

CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

• Parent, for Minor Patient

• Adult Patient or NIH-2514-1 (07-09)

P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study |
|---|---|
| | NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |

STUDY NUMBER: 09-C-0065 CONTINUATION:  pages

#### Why is this study being done?

Studies conducted at the National Cancer Institute suggest that certain chemotherapy drugs may be more effective if given by continuous infusion into the vein rather than by the standard method of rapid intravenous injection. One such combination, which we call EPOCH-R (each letter stands for one of the drugs used in the combination), seems to have a high degree of effectiveness in patients whose tumors have stopped responding to standard regimens. We therefore plan to test this combination in patients who have never received chemotherapy previously. Recent evidence also indicates that the effects of chemotherapy may be improved by combination with monoclonal antibodies. Monoclonal antibodies are purified proteins that are specially made to attach to pieces of foreign substances (such as cancer cells) with the goal of inactivating them. A monoclonal antibody, called siplizumab, has been manufactured to attach to a protein called CD2 that your type of tumor contains.

#### How many people will take part in this study?

Up to 30 patients will be treated on this study.

#### **Description of Research Study**

#### Objectives and design of this study:

The general purpose of this study is to develop treatments for lymphoma that are more effective than existing therapies. The experimental part of this treatment program is to test whether giving siplizumab in combination with continuous infusion EPOCH chemotherapy with filgrastim is safe and if it improves the outcome of therapy of your lymphoma. In this study five chemotherapy drugs are given together in an intensive combination called EPOCH. In addition, you will receive a drug called rituximab. Rituximab is another monoclonal antibody which binds to a specific molecule (called CD20) present on most B-cells. This drug is being given to help prevent a potential side effect of the siplizumab. EPOCH-R contains drugs which are standard for the treatment of lymphomas. Because higher doses of chemotherapy may increase the benefit, the doses of several drugs in EPOCH-R may be increased on each cycle if you tolerated them on the previous cycle.

#### Siplizumab-EPOCH-R chemotherapy treatment:

The chemotherapy regimen known as Siplizumab-EPOCH-R will be given by intravenous (IV) infusion through a "central line," an IV catheter (or tube) placed in a large vein in your arm or chest. You will be admitted to the hospital for the infusion of the monoclonal antibody therapy on this protocol but may receive the chemotherapy infusion as an outpatient. Patients will receive dose adjusted (DA) EPOCH-R chemotherapy which includes the following drugs: etoposide (E), prednisone (P), vincristine (O), cyclophosphamide (C), doxorubicin (H), and rituximab (R). The drug siplizumab will be given by IV infusion on the first day of treatment over several hours. When the siplizumab IV infusion is complete, the drugs doxorubicin, etoposide, and vincristine will each be given by continuous IV infusion over the next 4 days (that is, continuously for a total of 96 hours). When this infusion is completed, the drug rituximab will be given by IV infusion over several hours on Day 5. Cyclophosphamide will be given by IV infusion on Day 5.

#### PATIENT IDENTIFICATION

#### **CONTINUATION SHEET for either:**

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

MEDICAL RECORD

CONTINUATION SHEET for either:

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 09-C-0065 CONTINUATION:  pages

after you have received the previous chemotherapy drugs. Prednisone will be given by mouth (orally) twice each day for 5 days. You will take the first dose of prednisone 8-12 hours before starting the siplizumab.

You will receive the drug filgrastim by subcutaneous (under the skin) injection starting on Day 6 to increase white blood cell counts. Filgrastim will be continued until your white blood counts have reached acceptable levels. The dose of doxorubicin, etoposide, and/or cyclophosphamide may be "adjusted" up or down depending on your white blood cell count. You will be given a drug commonly known as Bactrim to be taken by mouth (orally) three times a week (for example, on a Monday-Wednesday-Friday schedule) to guard against possible infections. You will receive a drug called fluconazole to prevent fungal infections, and a drug called acyclovir to prevent certain viral infections. You will also receive a drug each day to be taken by mouth (orally) to guard against stomach ulcers, such as omeprazole. In addition, you will receive colace, or equivalent, by mouth twice daily to prevent constipation. If constipation becomes severe, you may also receive the laxative known as lactulose.

The siplizumab-EPOCH-R therapy will be repeated every twenty-one (21) days, which is known as a "cycle" of therapy, for a total of 6 cycles. Following the fourth and sixth treatment cycles (approximately weeks 12 and 18) of siplizumab- EPOCH-R, your doctor will evaluate you with blood tests and CT/MRI scans.

#### **Study Chart**

#### Siplizumab-EPOCH-R Treatment Schema

| | Dag | y of T | [reat | men | ıt | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | <br>21* |
| Siplizumab | | X | | | | | | | | | | | | | |
| Rituximab | | | | | | X | | | | | | | | | |
| Etoposide | | Х- | | - | - | <b>→</b> | | | | | | | | | |
| Prednisone | X | X | X | X | X | X | | | | | | | | | |
| Vincristine | | Х- | | - | - | <b>→</b> | | | | | | | | | |
| Cyclophosphamide | | | | | | X | | | | | | | | | |
| Doxorubicin | | X- | | | | $\rightarrow$ | | | | | | | | | |
| Filgrastim | | | | | | | X** | k | $\rightarrow$ | | | | | | |

<sup>\*</sup> This twenty-one day (21) period will be known as a "cycle" of therapy. Therapy will be repeated for a total of 6 cycles. During the course of treatment, you may also receive the following drugs:

PATIENT IDENTIFICATION

#### **CONTINUATION SHEET for either:**

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 09-C-0065 CONTINUATION:  pages

methotrexate, Bactrim, fluconazole, acyclovir, omeprazole, and colace. On the first cycle of therapy the start of EPOCH chemotherapy may be delayed until the following day if toxicity during the siplizumab infusion caused a prolonged infusion time.

\*\* Filgrastim will continue to be given to you until your blood counts have reached acceptable levels.

#### Treatment of disease in the nervous system:

Your lymphoma may spread to the central nervous system (CNS) which includes the brain and spinal cord. It may be necessary to treat the CNS with chemotherapy which usually includes the instillation of chemotherapy drugs (methotrexate and/or cytarabine) directly into the fluid (the cerebrospinal fluid, or CSF) surrounding the brain. This is usually done by first placing a small reservoir (called an Ommaya reservoir) under the skin of the scalp; this reservoir is connected to a catheter that is placed through the brain itself into the fluid. This procedure is performed by a neurosurgeon under general anesthesia. These drugs may also be administered through a spinal tap (also called a lumbar puncture). Depending on how you respond to this therapy, it may be necessary to modify it and/or to also administer radiation to your brain and/or spinal cord. Each of these therapies will be discussed with you if they are needed. Patients who have lymphoma in their bone marrow or in multiple areas outside of their lymph nodes are at higher risk of developing lymphoma in the brain areas. To reduce this risk, patients at higher risk will receive methotrexate by a spinal tap on day 1 of cycles 3-6 of their Siplizumab-EPOCH-R chemotherapy. Your treating physicians will discuss this with you.

#### Research tests:

We would like to perform research studies on your blood and tumor tissue to look at different genes and proteins that may be involved in the development of your lymphoma or the reaction of the immune system. We will not examine mutations of genes from your normal tissue without obtaining additional permission from you. We plan to do a tissue biopsy before you start treatment. Biopsies of tumor will be done with local or general anesthesia. The tumor biopsies are being performed for two reasons; first to confirm your diagnosis and test for CD2 and second to perform research tests on the tumor. These biopsies will give us important information about your tumor. Biopsies requiring major surgery (opening the chest or abdomen) will only be done if necessary for medical care and will not be done for experimental purposes. It is important, however, for you to understand that in some cases, biopsies of tumor may be done primarily for experimental purposes. These biopsies are optional for participation in the study but are important to help us learn how to better treat T cell lymphoma.

Certain patients who have tumor cells in their blood stream may be asked to undergo a procedure called lymphapheresis or apheresis for research purposes. Lymphapheresis or apheresis is done by circulating your blood through the apheresis machine. To do this you must have two places where IV needles are placed. There are two ways to do this procedure. In the first method, a needle is placed into each of your arm veins. The second method uses a vascular access device. Both methods provide a route for your blood to be circulated through the apheresis machine. Your blood is removed from one IV site, and then flows through the tubing into the machine. The machine has a centrifuge that separates the part of the blood that is to be removed. Only a

PATIENT IDENTIFICATION

#### **CONTINUATION SHEET for either:**

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consentto Participate in A Clinical Research Study |
|---|---|
| | NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |

STUDY NUMBER: 09-C-0065 CONTINUATION:  pages

small portion of your blood is circulated through the machine at any one time. The blood then returns to you through the other IV site. The procedure takes 2 - 4 hours to complete. Once the procedure is done, all of your blood is returned to you. You will be taken off the machine by the nurse. The needles are then removed and pressure is put over where the needles were to be sure that bleeding stops. After a period of rest, you will be told when to come in for your next procedure. The procedure may be done more than once.

Blood samples will be collected to measure the level of the siplizumab in your blood. During the first cycle, you will have ten samples drawn over a 5 day period. During cycles 2-6, you will only have 3 blood samples drawn. Each one of these samples will be slightly more than a teaspoon of blood.

You may have some discomfort when the nurse puts the needles into your veins. Keeping your arms in one position and staying still during a 2 - 4 hour procedure may also be a little uncomfortable. Some patients may feel dizzy, light-headed, nauseated, or cold during the procedure. Tell the staff right away if you feel any of these side effects. It is normal to feel tired for a short time after this procedure.

#### What happens after treatment is completed:

This depends on how you have responded to the therapy. If all evidence of disease has disappeared, we will schedule periodic visits to the Clinical Center for follow-up examination and tests. If the disease does not disappear entirely or if it should recur after having disappeared for a period of time, then you may need further therapy. At that time you will be given the opportunity of participating in additional research protocols that may be appropriate for you. If no such protocols are available, you will be returned to the care of your local physician. We will continue to contact you and/or your local physician to see how you are doing even after you have completed treatment on this protocol. It is important to stress that participation in this protocol does not constitute a promise of long-term medical care here at the Clinical Center. It is conceivable that participation in this study may make you ineligible to participate in certain other research protocols because the requirements for entry onto these protocols may not allow patients who have already been treated with certain drugs or who have had certain side effects from previous treatment. You may decide now not to receive treatment on this protocol, or you may choose at any point in time to stop the treatment and withdraw from the protocol; in either case you will be returned to the care of your referring physician.

#### Risks or Discomforts of Participation

In order to determine if you are eligible for this study, several tests need to be done. This period of evaluation may take up to three weeks and may be done on an outpatient basis. Evaluation may include some or all of the following tests: standard blood tests, 24 hour collections of urine, tests of lung and heart function, computerized tomography (CT) scans, nuclear medicine scans of the body (called a PET scan), bone marrow biopsies and biopsies of suspected areas of tumor.

PATIENT IDENTIFICATION

**CONTINUATION SHEET for either:** 

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consentto Participate in A Clinical Research Study |
|---|---|
| | NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |

STUDY NUMBER: 09-C-0065 CONTINUATION:  pages

The risks associated with bone marrow biopsies are pain, bleeding and local infection. Risks of tissue biopsies include pain, bleeding, infection, and the risks to the particular area undergoing surgery. A biopsy of tumor may require general anesthesia. General anesthesia itself is generally very safe but has a very small risk of major complications such as heart attack or stroke. The surgical and anesthetic risks will be explained to you in more detail at the time of surgery, if this is needed

You will undergo a lumbar puncture to remove a small amount of spinal fluid (about 1-2 teaspoons) that will be tested for the presence of lymphoma cells. A lumbar puncture is done by inserting a small sterile needle through the skin and muscle, going between the bones of the spine in the lower back until the needle punctures the spinal canal covering. The spinal fluid will then drain out through the needle on its own.

In order to receive this treatment, you will need to have a central venous catheter. This is catheter is placed under the skin of the chest wall and enters a major vein in the chest. There are several types of catheters including those which must be removed after each cycle of chemotherapy (temporary type) and those which may be kept for the duration of therapy (permanent type). These options will be discussed with you. The risks associated with placing some catheters include pain, bleeding, infection and collapsed lung. The long term risks of the catheter include infection, and clotting of your veins. If these occur, it may be necessary to remove the catheter. These risks will be explained to you in more detail at the time of insertion.

You may have side effects while on the study. Every one taking part in the study will be watched carefully for any side effects. However doctors don't know all the side effects that may happen. Side effects may be mild or serious. Your health care team may give you medicines to help lessen side effects. In some cases, side effects can be serious or long-lasting or may never go away. There is also the risk of death from either the treatment or your disease.

You should talk to your doctor about any side effects that you have while taking part in the study. Risks and side effects related to the treatment are identified below.

#### **Side Effects of Siplizumab:**

"Likely" side effects occur in greater than 50% of patients. "Less likely" side effects occur in 10-50% of patients. "Occasional" side effects occur in <10% of patients. "Unlikely" side effects occur in <1% of patients. "Serious" side effects are severe, life threatening, or cause death. Most of the side effects are listed in this form, but they will vary from person to person. There may be other side effects that we don't know about.

#### Likely:

• Mild flu-like symptoms such as chills, fever (usually occur only with the first dose and decreased or absent with each following dose). Stopping or increasing the time it takes to give you siplizumab may make these side effects go away.

PATIENT IDENTIFICATION

**CONTINUATION SHEET for either:** 

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study |
|---|---|
| | NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |

STUDY NUMBER: 09-C-0065 CONTINUATION:  pages

Decreased white blood cells (including normal T-cells), which may increase the risk of
infection (bacterial, viral, fungal, parasitic); you will be given medicines to prevent
infections.

**Less likely-**-these usually occur only with the first dose and are decreased or absent with each following dose:

- Dizziness
- nausea
- general sick feeling
- muscle pain
- headache

#### Occasional:

- Anemia (decreased red blood cells, which causes you to feel tired, lightheaded, and have a rapid heartbeat)
- anorexia (lack of appetite)
- diarrhea
- cold sores (herpes simplex)
- high or low blood pressure
- paresthesia (abnormal touch sensation)
- sore throat
- itching
- rapid or slow heart beat
- sweating
- abnormal taste
- vasodilatation (increased blood flow)
- weakness

#### Unlikely:

- Ecchymosis (small hemorrhagic spot in the skin)
- hyperesthesia (increased pain sensitivity)
- hypothermia (low body temperature)
- difficulty sleeping
- leg cramps
- leukocytosis (temporary increase in white blood cells)
- pain

### PATIENT IDENTIFICATION CONTINUATION SHEET for either: NIH-2514-1 (07-09) NIH-2514-2 (10-84)

P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 09-C-0065 CONTINUATION:  pages

- pleural (lining of the lung) disorder
- decrease in platelets

#### Unlikely, but serious:

- Allergic reactions with any of the following symptoms:
  - Marked lowering of the blood pressure, throat tightness, shortness of breath, severe skin rash
- Development of other cancers or recurrence of a past cancer.
- Development of Epstein-Barr Virus associated disease that may be malignant (up to about 10% of patients treated with siplizumab.
- Shock-like reaction, which may include heart, lung, and brain problems, caused by the killing of normal T-cells.
- Heart rhythm, kidney, and lung problems caused by chemicals released into your blood from dead cancer cells; you will receive extra fluids before you start your treatment with siplizumab to flush any extra chemicals out of your body, and you will also be given medicine to help control the chemical balance of your blood.
- Inflammation of the joints
- Serious viral infection
- Changes in liver enzymes

Since siplizumab can cause a prolonged lowering of lymphocytes (white blood cells), you may develop an increased risk for serious infections, the development of other tumors, or the recurrence of a previous cancer. Also, it is important to know that patients may develop other unexpected side effects and these could lead to serious organ damage or even death.

#### **Side Effects of EPOCH-R:**

#### Likely:

- Lowered white blood cell count that may lead to infection
- Lowered platelets which may lead to an increase in bruising or bleeding
- Lowered red blood cells which may cause anemia, tiredness, or shortness of breath
- Should low counts occur, they can be treated with blood products (transfusions), antibiotics, and there may be a reduction in the amount of drug given to you
- Constipation
- Fatigue or tiredness
- Tingling of fingers and/or toes
- Hair loss

| PATIENT IDENTIFICATION | CONTINUATION SHEET for either: |
|------------------------|-------------------------------------|
| | NIH-2514-1 (07-09) |
| | NIH-2514-2 (10-84) |
| | P.A.: 09-25-0099 |
| | File in Section 4: Protocol Consent |

## MEDICAL RECORD CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 09-C-0065 CONTINUATION:  pages

- Fever and/or chills
- Time away from work
- Urine colored red for a day or two after the doxorubicin infusion
- Fingernail and toenail changes
- Tearing or dry eyes
- Runny nose
- Bony pain

#### Less Likely:

- Nausea and/or vomiting
- Loss of appetite, change in taste and weight loss
- Temporary shortness of breath or dizziness while receiving rituximab
- Headaches
- Muscle aches and muscle weakness
- Hoarseness or pain in the jaw
- Elevated blood sugar levels
- Elevated or decreased blood pressure
- Confusion
- Mouth & throat sores. Temporary irritation to the mouth may lead to mouth ulcers (similar to canker sores). Medications to numb the mouth may ease the mouth discomfort.
- Stomach ulcers
- Skin rashes and/or dry skin
- Loss of control of muscles or reflexes
- Abnormalities in blood results such as elevated liver enzymes, low blood protein and low blood calcium
- Mood changes such as agitation or depression
- Trouble sleeping

#### Rare, But Serious:

- Severe constipation may result in abdominal pain and cramping
- Bladder irritation with painful and bloody urine
- Damage to the heart muscle
- Skin rash that may be serious and life-threatening
- Allergic reaction that may be severe or life-threatening. Symptoms may include difficulty breathing, low blood pressure, fast heart rate, and sweating.

# PATIENT IDENTIFICATION CONTINUATION SHEET for either: NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099 File in Section 4: Protocol Consent

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 09-C-0065 CONTINUATION:  pages

• Severe hepatitis (liver infection) in those patients who are carriers of the hepatitis virus. Patients who may have had prior exposure to the hepatitis B and C virus may be at an increased risk of recurrence of the virus that may lead to severe liver damage that can be life-threatening. You doctor will screen you for the hepatitis virus before beginning treatment on this study. If you test positive for the virus, you will be closely monitored for signs of the infection, and you will be treated, if appropriate, by your doctor.

#### Drugs used for the treatment of the nervous system:

- Methotrexate, when administered into the spinal fluid, may cause low blood counts and ulcerations in the mouth, stomach, and intestines. It can cause acute headache, back pain, stiff neck, and /or fever; it can also cause weakness or paralysis of certain muscles. It can cause seizures and coma. Other side effects it can cause are usually associated with intravenous administration rather than intrathecal (lumbar puncture administration), but these include liver function abnormalities, inflammation and scarring of the lungs, inflammation of the tissue covering the heart, and severe skin reactions.
- Cytarabine given by lumber puncture can cause nausea, vomiting, fever, and headaches. Rarely, it can cause weakness and seizures. When given into the spinal fluid, it does not usually cause systemic toxicity, but we will monitor you for low blood counts, and liver function abnormalities, which can occur with cytarabine when given by vein.

#### **Secondary Malignancy:**

A number of established chemotherapy agents have an inherent risk of causing another cancer (known as a "secondary malignancy"). Certain drugs in use today, not currently known to be associated with this risk may be shown at a later time to result in the development of these secondary malignancies. Siplizumab, when used by itself, has rarely caused a secondary cancer related to the Epstein-Barr virus (EBV). The rituximab is given in this regimen to help prevent this. If you do develop an EBV related cancer, you will not receive any more siplizumab therapy. The treatment of EBV related cancer ranges from observation to treatment with rituximab alone or with chemotherapy.

#### **Reproductive Risks:**

Many of the drugs used in this treatment program are toxic to the cells in the ovary and testicle and may produce sterility. Recovery of normal fertility is not well studied although we know that some patients treated with this combination have remained fertile after the therapy has been completed. For this reason, men who are about to receive this treatment should, if they wish to have children in the future, consider sperm banking before start of the treatment. These drugs, as well as the scans performed to assess your disease may also be very toxic to an unborn child or nursing baby. Therefore, adequate birth control measures (such as the contraceptive pill, condoms, diaphragm with contraceptive foam or ointment, contraceptive sponge, etc.) should be used by participants or their sexual partners while receiving treatment on this study. Women of childbearing age will have a pregnancy test, which must be negative at the time of study entry. This test requires that blood be drawn from a vein one or two days prior to the study. The results

PATIENT IDENTIFICATION

#### **CONTINUATION SHEET for either:**

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| CONTINUATION SHEET for either: NIH 2514-1, Consentto Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|
|---|

STUDY NUMBER: 09-C-0065 CONTINUATION:  pages

of the pregnancy test will be made available to you prior to the initiation of the study. If you are a woman and become pregnant while on this study, treatment will be stopped. If you think that you may have become pregnant while you are on this study, please contact the Principal Investigator, Dr. Wyndham Wilson, Telephone: 240-760-6092, before taking any further study treatment or undergoing any imaging scans.

#### **Infection Risks:**

It is important to emphasize that when you have a decreased white blood cell count you are at risk of infection. Such infections can be very serious and can even cause death if not quickly and properly treated. If you have a temperature greater than 38.3° C (101° F), you must call your doctor immediately. If your temperature is higher than 38.0° C (100.4° F) two times in a 24 hour period, you must call your doctor immediately. Chemotherapy may also cause your platelets to fall; since platelets are the blood elements that permit blood to clot, this may place you at increased risk of serious bleeding. It may be necessary to give you transfusions of platelets if your platelet counts reach very low levels. There is a small chance that damage to the normal bone marrow may eventually result in bone marrow failure, leading to a serious shortage of one or more kinds of cells in the blood, or to leukemia.

Your physicians will watch you closely for side effects and will stop treatment if any side effects become a serious threat to your life or well-being. Your physicians will also stop the treatments if it becomes clear that the treatment is not successfully controlling your disease. For more information about risks and side effects, ask your study doctor.

#### Risks of Treatment of the Central Nervous System:

It may be necessary to treat the CNS with chemotherapy which usually includes the instillation of chemotherapy drugs (methotrexate and/or cytarabine) directly into the fluid (the cerebrospinal fluid, or CSF) surrounding the brain. This is usually done by first placing a small reservoir (called an Ommaya reservoir) under the skin of the scalp; this reservoir is connected to a catheter that is placed through the brain itself into the fluid. Complications of Ommaya insertion are uncommon when done by an experienced doctor but could include infection and bleeding at the operative site or in the brain itself. Complications of lumbar puncture may include pain or bleeding at the site of needle insertion (the low back), infection, and headache. Most patients tolerate this treatment without serious side effects, although drugs placed into the brain fluid (CSF) may cause headache, stiff neck, and confusion that resolve when they are stopped. With long-term treatment, confusion and a slowing of thought processes may occur. If this treatment becomes necessary for you, the complications of the lumbar puncture or Ommaya insertion and methotrexate instillation will be discussed in more detail.

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consentto Participate in A Clinical Research Study |
|---|---|
| | NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |

STUDY NUMBER: 09-C-0065

CONTINUATION:  pages

#### Potential Benefits of Participation

#### Are there benefits to taking part in this study?

It is likely that most patients will have at least a temporary improvement from treatment with Siplizumab and EPOCH-R chemotherapy. However, we cannot be certain if you will be cured of your lymphoma and it is possible that you may not respond to treatment.

In addition, your participation in this protocol may contribute to advances in the understanding of and treatment for your disease.

#### **Alternative Approached or Treatments**

#### What other choices do I have if I do not take part in this study?

It should be emphasized that we do not know at this point whether the combination of drugs we propose to give you is superior, inferior or equivalent to standard combination chemotherapy for your disease. Alternative procedures that could be used to treat your disease include:

- Other combination drug regimens and other schedules of the same drugs used in this study. For example, a chemotherapy called CHOP given in the conventional manner would be suitable standard therapy for your condition.
- Treatment with single drugs. This is known to produce brief responses of a few months'
  duration in many patients but to have little beneficial effect in long-term control of the
  disease.
- Radiation (X-ray) treatments. This can stop tumor growth in particular locations, such as bone, abdomen, and other sites but is not successful in controlling the disease overall unless the disease is very localized at the start of therapy.
- Surgery. As with radiation, surgery can be successful in removing tumor from particular
  locations but cannot be used successfully to remove all lymphoma cells from the body,
  since the disease is almost always present in multiple locations. Also, surgery cannot be
  used against tumor in some of the organs most commonly involved by lymphoma, such
  as the liver or the lungs.
- Waiting, without active therapy. Although a period of watchful waiting is appropriate treatment for some kinds of tumors, in lymphomas similar to yours, the disease will often grow and spread rapidly if no treatment is administered.
- No treatment. You can choose not to receive any therapy for your lymphoma. In this case, your doctor can give you medications that will make you feel comfortable.

#### **Stopping Therapy**

Your doctor may decide to stop your therapy for the following reasons:

- if he/she believes that it is in your best interest
- if your disease comes back during treatment

## PATIENT IDENTIFICATION CONTINUATION SHEET for either: NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099 File in Section 4: Protocol Consent

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consentto Participate in A Clinical Research Study |
|---|---|
| | NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |

STUDY NUMBER: 09-C-0065 CONTINUATION:  pages

- if you have side effects from the treatment that your doctor thinks are too severe
- if new information shows that another treatment would be better for you

In this case, you will be informed of the reason therapy is being stopped.

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. However, according to FDA guidelines, information collected on you up to that point may still be provided to MedImmune or designated representatives. If you withdraw your consent and leave the trial, any samples of yours that have been obtained for the study and stored at the NCI can be destroyed upon request. However, any samples and data generated from the samples that have already been distributed to other researchers or placed in the research databases can**not** be recalled and destroyed.

#### Research Subject's Rights

#### What are the costs of taking part in this study?

If you choose to take part in the study, the following will apply, in keeping with the NIH policy:

- You will receive study treatment at no charge to you. This may include surgery, medicines, laboratory testing, x-rays or scans done at the Clinical Center, National Institutes of Health (NIH), or arranged for you by the research team to be done outside the Clinical Center, NIH if the study related treatment is not available at the NIH.
- There are limited funds available to cover the cost of some tests and procedures performed outside the Clinical Center, NIH. You may have to pay for these costs if they are not covered by your insurance company.
- Medicines that are not part of the study treatment will not be provided or paid for by the Clinical Center, NIH.
- Once you have completed taking part in the study, medical care will no longer be provided by the Clinical Center, NIH.

#### Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The National Cancer Institute (NCI) and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Institutes of Health Intramural Institutional Review Board
- The study Sponsor (Medimmune)
- Qualified representatives from Medimmune, the pharmaceutical company who produces siplizumab.

| 1 | |
|------------------------|-------------------------------------|
| PATIENT IDENTIFICATION | CONTINUATION SHEET for either: |
| | NIH-2514-1 (07-09) |
| | NIH-2514-2 (10-84) |
| | P.A.: 09-25-0099 |
| | File in Section A: Protocol Consent |

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 09-C-0065 CONTINUATION:  pages

A description of this clinical trial will be available on <a href="http://www.Clinicaltrials.gov">http://www.Clinicaltrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most the Web site will include a summary of the results. You can search this Web site at any time.

#### **Certificate of Confidentiality**

To help us protect your privacy, we have obtained a Certificate of Confidentiality. The researchers can use this Certificate to legally refuse to disclose information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if there is a court subpoena. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below.

You should also know that there are several circumstances in which the Certificate does not provide coverage. These include when information:

- will be used for auditing or program evaluation internally by the NIH; or
- must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA).
- is necessary for your medical treatment and you have consented to this disclosure;
- is for other research.

In addition, identifiable, sensitive information protected by this Certificate cannot be admissible as evidence or used for any purpose in any action, suit, or proceeding without your consent.

You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then the researchers will not use the Certificate to withhold that information.

The Certificate of Confidentiality will not protect against the required reporting by hospital staff of information on suspected child abuse, reportable communicable diseases, and/or possible threat of harm to self or others.

#### **Conflict of Interest**

The National Institutes of Health (NIH) reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a Protocol Review Guide. You may ask your research team for a copy of the Protocol Review Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines but they do not need to report their personal finances to the NIH.

Members of the research team working on this study may have up to \$15,000 of stock in the manufacturer of the product(s) used in this study. This is allowed under federal rules and is not a conflict of interest.

NIH-2514-1 (07-09) NIH-2514-2 (10-84)

P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 09-C-0065 CONTINUATION:  pages

• The National Institutes of Health and the research team for this study are using siplizumab developed by MedImmune, Inc. through a joint study with your researchers and the company. The company also provides financial support for this study.

#### Use of Specimens and Data for Future Research

To advance science, it is helpful for researchers to share information they get from studying human samples. They do this by putting it into one or more scientific databases, where it is stored along with information from other studies. A researcher who wants to study the information must apply to the database and be approved. Researchers use specimens and data stored in scientific databases to advance science and learn about health and disease.

We plan to keep some of your specimens and data that we collect and use them for future research and share them with other researchers. We will not contact you to ask about each of these future uses. These specimens and data will be stripped of identifiers such as name, address or account number, so that they may be used for future research on any topic and shared broadly for research purposes. Your specimens and data will be used for research purposes only and will not benefit you. It is also possible that the stored specimens and data may never be used. Results of research done on your specimens and data will not be available to you or your doctor. It might help people who have cancer and other diseases in the future.

If you do not want your stored specimens and data used for future research, please contact us in writing and let us know that you do not want us to use your specimens and/or data. Then any specimens that have not already been used or shared will be destroyed and your data will not be used for future research. However, it may not be possible to withdraw or delete materials or data once they have been shared with other researchers.

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

#### MEDICAL RECORD

#### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

Adult Patient or

• Parent, for Minor Patient

STUDY NUMBER: 09-C-0065

CONTINUATION:  pages

#### OTHER PERTINENT INFORMATION

1. Confidentiality. When results of an NIH research study are reported in medical journals or at scientific meetings, the people who take part are not named and identified. In most cases, the NIH will not release any information about your research involvement without your written permission. However, if you sign a release of information form, for example, for an insurance company, the NIH will give the insurance company information from your medical record. This information might affect (either favorably or unfavorably) the willingness of the insurance company to sell you insurance.

The Federal Privacy Act protects the confidentiality of your NIH medical records. However, you should know that the Act allows release of some information from your medical record without your permission, for example, if it is required by the Food and Drug Administration (FDA), members of Congress, law enforcement officials, or authorized hospital accreditation organizations.

- 2. Policy Regarding Research-Related Injuries. The Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the National Institutes of Health, the Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.
- **3. Payments.** The amount of payment to research volunteers is guided by the National Institutes of Health policies. In general, patients are not paid for taking part in research studies at the National Institutes of Health. Reimbursement of travel and subsistence will be offered consistent with NIH guidelines.
- **4. Problems or Questions.** If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Wyndham Wilson, M.D., Ph.D.; Building 10, Room 4N115, Telephone: 240-760-6092. You may also call the Clinical Center Patient Representative at (301) 496-2626. If you have any questions about the use of your specimens or data for future research studies, you may also contact the Office of the Clinical Director, Telephone: 240-760-6070.
- 5. Consent Document. Please keep a copy of this document in case you want to read it again.

PATIENT IDENTIFICATION

**CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY (Continuation Sheet)** 

• Adult Patient or NIH-2514-1 (07-09)

• Parent, for Minor Patient

P.A.: 09-25-0099

MEDICAL RECORD

#### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

Adult Patient or

• Parent, for Minor Patient

STUDY NUMBER: 09-C-0065

CONTINUATION:  pages

| COMPLETE APPROPRIATE ITEM(S) BELOW: | | | |
|---|---|---|---|
| A. Adult Patient's Consent | | B. Parent's Permission for Minor Patient. | |
| I have read the explanation about this study<br>and have been given the opportunity to discuss<br>it and to ask questions. I hereby consent to<br>take part in this study. | | I have read the explanation about this study<br>and have been given the opportunity to discuss<br>it and to ask questions. I hereby give<br>permission for my child to take part in this<br>study. | |
| | | (Attach NIH 2514-2, Minor's Asso<br>applicable.) | ent, if |
| Signature of Adult Patient/ Legal Representative | Date | Signature of Parent(s)/ Guardian | Date |
| Legal Representative | | | |
| Print Name | | Print Name | |
| C. Child's Verbal Assent (If Appl<br>The information in the above consen<br>participate in the study. | | bed to my child and my child agree | s to |
| Signature of Parent(s)/Guardian | Date | Print Name | |
| THIS CONSENT DOCUMENT HAS BEEN APPROVED FOR USE FROM FEBRUARY 5, 2018 THROUGH FEBRUARY 4, 2019. | | | |
| Signature of Investigator | Date | Signature of Witness | Date |
| Print Name | | Print Name | |

PATIENT IDENTIFICATION

### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY (Continuation Sheet)

• Adult Patient or NIH-2514-1 (07-09) • Parent, for Minor Patient

P.A.: 09-25-0099